CLINICAL TRIAL: NCT06994741
Title: Retrospective Study of Gait Parameters in a Cohort of Patients Fitted With a Canadian Prosthesis: Contribution of Quantified Gait Analysis
Brief Title: Gait Parameters in a Cohort of Patients Fitted With a Canadian Prosthesis: Contribution of Quantified Gait Analysis
Status: Completed | Type: Observational
Sponsor: Institut Robert Merle d'aubigné (Other)
Responsible Party: Sponsor
Other Study IDs: 2024 - RNIPH - 001
Record Dates: First submitted 2025-04-15; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Amputation; Gait, Unsteady
Keywords: Canadian prothesis
MeSH Terms: conditions — Gait Disorders, Neurologic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Amputee with canadian prothesis
  Interventions: Other: Quantitative movement analysis

INTERVENTIONS:
Other: Quantitative movement analysis — During their reeducation, patient can go through an quantitative movement analysis. Inside a movement laboratory, we observe their gait with 5 passageways.

SUMMARY:
The goal of this clinical trial is to learn about the biomechanics characterics of amputee with a canadian prothesis during gait. The main question to answer is : what are the main biomechanical characteristics and their statistical description.

Participant had pass through a quantitative movement analysis during their classic reeducaiton and we are going to use these data.

ELIGIBILITY:
Inclusion Criteria:

* with canadian prothesis
* presence of the gait analysis

Exclusion Criteria:

* major gait disorder due to another pathologie
* major gait disorder due to a wrong adapration of the prothesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: amputee with canadian prothesis
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Walking speed | Day 1
  (m/s) with a motion laboratory - Vicon system with 8 cameras, Nexus 2.4 et Polygon 2.4

SECONDARY OUTCOMES:
Joint range of motion | Day 1
  (°) with a motion laboratory - Vicon system with 8 cameras, Nexus 2.4 et Polygon 2.4
Force apply to the ground | Day 1
  (N/m2) with a motion laboratory and 2 forceplates AMTI - Vicon system with 8 cameras, Nexus 2.4 et Polygon 2.4
Steplength | During the quantitative movement analysis - retrospective data

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Robert Merle d'Aubigné, Valenton, Val-de-Marne, France

IPD SHARING:
Plan to Share IPD: Undecided